CLINICAL TRIAL: NCT01193556
Title: A Prospective, Randomized, Double-blinded, Controlled Study to Evaluate Use of the PEAK PlasmaBlade TnA in Subcapsular Tonsillectomy
Brief Title: PEAK PlasmaBlade TnA Versus Traditional Electrosurgery in Subcapsular Tonsillectomy
Acronym: PRECISE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Termination due to acquisition of PEAK Surgical by Medtronic
Sponsor: Medtronic Surgical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEAK VP-00075
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Results first posted 2013-01-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-11

CONDITIONS: Tonsillitis
Keywords: Tonsillectomy; PlasmaBlade; Electrosurgery; PEAK Surgical; Medtronic Advanced Energy; Medtronic
MeSH Terms: conditions — Tonsillitis; Hyperthermia | interventions — Electrosurgery; Electrocoagulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Active Comparator): Traditional electrosurgery will be used for the tonsillectomy.
  Interventions: Device: Traditional Electrosurgery with scalpel
- PlasmaBlade (Experimental): The PEAK PlasmaBlade will be used for the tonsillectomy.
  Interventions: Device: PEAK PlasmaBlade TnA

INTERVENTIONS:
Device: PEAK PlasmaBlade TnA — The PEAK PlasmaBlade will be used for the tonsillectomy.
  Other Names: PEAK; PlasmaBlade; Plasma Blade; TnA; Tonsil and Adenoid
  Arms: PlasmaBlade
Device: Traditional Electrosurgery with scalpel — Traditional electrosurgery for the tonsillectomy.
  Other Names: Electrosurgery; Electrocautery; Bovie
  Arms: Standard of Care

SUMMARY:
The objective of this clinical study is to evaluate the operative performance of the PEAK PlasmaBlade® TnA during subcapsular tonsillectomy; to monitor and record post-operative clinical outcome variables; and to compare these endpoints to the Standard of Care (SOC).

DETAILED DESCRIPTION:
Tonsillectomy is performed in response to cases of repeated occurrence of acute tonsillitis or adenoiditis, obstructive sleep apnea, nasal airway obstruction, snoring, or peritonsillar abscess.

The PEAK PlasmaBlade uses pulsed radiofrequency (RF) energy and a highly-insulated handpiece design to enable precision cutting and coagulation at the point of application. The PlasmaBlade has received FDA clearance for use in plastic, general, orthopedic, and ear, nose, and throat (ENT) surgery, and has demonstrated a significantly reduced thermal injury profile in incised tissue compared to traditional electrosurgical devices. It is hypothesized that this benefit may improve the post-operative outcome of patients undergoing tonsillectomy.

Two study sites were granted approval for this prospective randomized study. Potential subjects were screened against the inclusion and exclusion criteria of the study protocol and were required to provide informed consent for themselves (adults) or for their child prior to enrollment. Following enrollment, subjects were prospectively randomized to the SOC or PlasmaBlade (PB or PEAK) study groups and scheduled for tonsillectomy or tonsillectomy and adenoidectomy (TnA).

ELIGIBILITY:
Inclusion Criteria:

1. Children & adolescents: Age 3-17; Adults: 18 and older
2. Physically healthy, stable weight
3. Requiring tonsillectomy and adenoidectomy per widely accepted indications
4. For adults, subject must understand the nature of the procedure and provide written informed consent.
5. For children and adolescents age 7 to 17, subject must understand the nature of the procedure and be able to give verbal assent prior to the procedure. In addition, parent or guardian must provide written informed consent.
6. For children under 7 years old, parent or guardian must understand the nature of the procedure and provide written informed consent.
7. Subject (or responsible parent or guardian) must be willing and able to comply with all follow-up evaluations, including completion of study data sheets.

Exclusion Criteria:

1. Children: Age 2 and under
2. Bleeding disorder
3. Peritonsillar abscess
4. Requiring concomitant uvulopalatopharyngoplasty (UPPP)
5. Anticoagulation therapy which cannot be discontinued
6. Unable to follow instructions or complete follow-up
7. Currently taking any medication known to affect healing
8. Currently enrolled in another investigational device or drug trial

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-07; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Weeks, MD, Principal Investigator — Senta Clinic; Mark Spitzer, DO, Principal Investigator — Mark Spitzer, DO
Locations (2):
- United States (2):
  - University Surgery Center Merced, Merced, California
  - Alvarado Hospital, San Diego, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care (SOC): Traditional electrosurgery will be used for the tonsillectomy.
Period: Overall Study
Arm/Group | Standard of Care (SOC) | PlasmaBlade
Started | 26 | 25
Completed | 0 | 0
Not Completed | 26 | 25
Not completed — Study termination | 26 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SOC) | PlasmaBlade | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Customized [Number; unit: participants]
  Children (3-17 years) | 14 | 13 | 27
  Adults (18 years and older) | 12 | 12 | 24
Gender [Number; unit: partipants]
  Female | NA — An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation. | NA — An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation. | 0
  Male | NA — An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation. | NA — An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation. | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain
Description: The primary outcome measure will be pain in each treatment group, as measured by visual analog scale twice daily in the 10 day period directly following surgery.
Time Frame: 10 days immediately following surgery
Population: An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation.
Arm/Group | Standard of Care (SOC) | PlasmaBlade
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Operative Time, Estimated Blood Loss (EBL), Diet Volume and Activity Level
Time Frame: 1-2 weeks post-operatively
Population: An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation.
Arm/Group | Standard of Care (SOC) | PlasmaBlade
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Standard of Care (SOC) | PlasmaBlade
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/25
Other Adverse Events (participants affected / at risk) | 0/26 | 4/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SOC) (N=26) | PlasmaBlade (N=25)
Postoperative bleeding (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SOC) (N=26) | PlasmaBlade (N=25)
Nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Postoperative bleeding (Surgical and medical procedures) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Upon Medtronic's acquisition of PEAK surgical, a study integrity audit was undertaken. Results of the audit showed that patient's rights and safety were maintained, but the source data, including baseline demographics, were unverifiable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less